CLINICAL TRIAL: NCT04732143
Title: The Effect of Preoperative Inspiratory Muscle Training Using Incentive Spirometer on Postoperative Pulmonary Complications Following Lung Resection
Brief Title: Effect of Preoperative Incentive Spirometer on Postoperative Pulmonary Complications Following Lung Resection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and clinical resources to continue
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Pauline Go, Associate Professor of Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00015501
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Respiratory Complication
Keywords: Incentive Spirometry; Inspiratory Muscle Training; Pulmonary Resection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive Spirometry (Experimental): Participants will undergo inspiratory muscle training using an incentive spirometer daily for 14 days prior to surgery.
  Interventions: Other: Inspiratory muscle training
- Standard Care (No Intervention): Participants will not undergo any inspiratory muscle training prior to surgery.

INTERVENTIONS:
Other: Inspiratory muscle training — At least 2 weeks prior to surgery, participants will be given a Vyaire incentive spirometer device and provided with formal training on proper inspiratory muscle breathing exercise using the device. They will be instructed to perform 4 sets of these exercises per day for 14 days prior to surgery.
  Other Names: Incentive spirometry
  Arms: Incentive Spirometry

SUMMARY:
The objective of this study is to demonstrate that inspiratory muscle training with daily use of an incentive spirometer for at least 14 days prior to lung surgery will reduce the risk of post-operative pulmonary complications.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPC) are the most common adverse events following lung resection, with a reported incidence of over 20-30% in some series. The objective of this study is to demonstrate that inspiratory muscle training (IMT) with daily use of an incentive spirometer (IS) for at least 14 days prior to lung surgery will reduce the risk of PPCs compared to the usual care, consisting of no formal preoperative IMT. The hypothesis is that preoperative inspiratory spirometer breathing (ISB) is a feasible and cost-effective intervention that can significantly reduce PPCs after lung resection. It is also hypothesized that patient compliance with the intervention will be high because of its simplicity, convenience, low cost and no potential for adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status score 2 or less
* Undergoing elective lung resection (includes wedge resection, lobectomy, bi-lobectomy, pneumonectomy, sleeve resection) via minimally invasive (VATS or robotic) approach or thoracotomy
* Chest wall resection if performed concurrently with lung resection

Exclusion Criteria:

* ECOG performance status score greater than 2
* Significant cognitive impairment preventing informed consent
* Non-English speaking
* Wedge biopsy for interstitial lung disease
* Bullectomy for bullous emphysema
* Pre-existing tracheostomy
* Emergent or urgent surgery
* Preoperative home oxygen use
* History of neuromuscular disease
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Atelectasis | Through completion of follow-up (30 days)
  Incidence of atelectasis requiring bronchoscopy or additional bedside therapy by a respiratory therapist
Pneumonia | Through completion of follow-up (30 days)
  Clinical and/or radiographic evidence of pneumonia requiring antibiotic therapy
Respiratory failure | Through completion of follow-up (30 days)
  Incidence of respiratory failure requiring re-intubation or high flow nasal cannula and/or non-invasive positive pressure ventilation
Pleural effusion | Through completion of follow-up (30 days)
  Incidence of pleural effusion requiring drainage or other medical intervention (e.g. use of diuretics)
Pneumothorax or subcutaneous emphysema | Through completion of follow-up (30 days)
  Incidence of clinically significant pneumothorax or subcutaneous emphysema requiring intervention or extended hospital admission for observation
Prolonged air leak | Through completion of follow-up (30 days)
  Incidence of prolonged air leak (>5 days) or requiring discharge with chest tube
Need for supplemental oxygen | Through completion of follow-up (30 days)
  Incidence of patients requiring supplemental oxygen upon discharge
Empyema/bronchopleural fistula | Through completion of follow-up (30 days)
  Incidence of empyema and/or bronchopleural fistula confirmed by fluid analysis and/or cultures
Cardiac arrhythmia | Through completion of follow-up (30 days)
  Incidence of cardiac arrhythmia requiring intervention (e.g. atrial fibrillation, supraventricular tachycardia, etc.)

SECONDARY OUTCOMES:
Hospital length of stay | Through completion of follow-up (30 days)
  Total length of index admission following surgery
ICU length of stay | Through completion of follow-up (30 days)
  If participant required ICU admission
Chest tube duration | Through completion of follow-up (30 days)
  Number of days from chest tube insertion (surgery date) until chest tube removal
Hospital readmission | Through completion of follow-up (30 days)
  Participant visited an emergency department and/or was admitted to the hospital following discharge from the index admission for any reason.
Change from baseline in dyspnea, measured by the modified Medical Research Council scale | Baseline, 2 weeks and 4 weeks after surgery
  Scores are measured on a scale from 0 to 4, with 0 indicating dyspnea only with strenuous exercise and 4 indicating participant is too dyspneic to leave the house or breathless when dressing
Mortality | Through completion of follow-up (30 days)
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pauline H Go, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Pehlivan E, Turna A, Gurses A, Gurses HN. The effects of preoperative short-term intense physical therapy in lung cancer patients: a randomized controlled trial. Ann Thorac Cardiovasc Surg. 2011;17(5):461-8. doi: 10.5761/atcs.oa.11.01663. Epub 2011 Jul 13. PMID 21881371
- [Background] Gao K, Yu PM, Su JH, He CQ, Liu LX, Zhou YB, Pu Q, Che GW. Cardiopulmonary exercise testing screening and pre-operative pulmonary rehabilitation reduce postoperative complications and improve fast-track recovery after lung cancer surgery: A study for 342 cases. Thorac Cancer. 2015 Jul;6(4):443-9. doi: 10.1111/1759-7714.12199. Epub 2014 Dec 22. PMID 26273399
- [Background] Valkenet K, Trappenburg JCA, Ruurda JP, Guinan EM, Reynolds JV, Nafteux P, Fontaine M, Rodrigo HE, van der Peet DL, Hania SW, Sosef MN, Willms J, Rosman C, Pieters H, Scheepers JJG, Faber T, Kouwenhoven EA, Tinselboer M, Rasanen J, Ryynanen H, Gosselink R, van Hillegersberg R, Backx FJG. Multicentre randomized clinical trial of inspiratory muscle training versus usual care before surgery for oesophageal cancer. Br J Surg. 2018 Apr;105(5):502-511. doi: 10.1002/bjs.10803. PMID 29603130
- [Background] Weiner P, Man A, Weiner M, Rabner M, Waizman J, Magadle R, Zamir D, Greiff Y. The effect of incentive spirometry and inspiratory muscle training on pulmonary function after lung resection. J Thorac Cardiovasc Surg. 1997 Mar;113(3):552-7. doi: 10.1016/S0022-5223(97)70370-2. PMID 9081102
- [Background] Benzo R, Wigle D, Novotny P, Wetzstein M, Nichols F, Shen RK, Cassivi S, Deschamps C. Preoperative pulmonary rehabilitation before lung cancer resection: results from two randomized studies. Lung Cancer. 2011 Dec;74(3):441-5. doi: 10.1016/j.lungcan.2011.05.011. Epub 2011 Jun 12. PMID 21663994